CLINICAL TRIAL: NCT03025997
Title: The Effect of Orally Applied Encapsulated Lipids in Yoghurt on Satiety and Food Intake: a Randomized Single-blind Placebo-controlled Study With Cross-over Design
Brief Title: Lipid Encapsulation for Ileal Brake Activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Wageningen University and Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: NL59245.068.16; 163042 (Other: METC)
Record Dates: First submitted 2017-01-06; First posted 2017-01-20 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-03

CONDITIONS: Appetite Regulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active yoghurt (Active Comparator): Yoghurt snack containing encapsulated lipid
  Interventions: Dietary Supplement: Active yoghurt
- Placebo yoghurt (Placebo Comparator): Yoghurt snack containing non-encapsulated lipid
  + empty encapsulation matrix
  Interventions: Dietary Supplement: Placebo yoghurt

INTERVENTIONS:
Dietary Supplement: Active yoghurt — Active yoghurt (containing encapsulated lipid) will be ingested after a standardized breakfast, and subsequently satiety and food intake will be measured.
  Arms: Active yoghurt
Dietary Supplement: Placebo yoghurt — Placebo yoghurt (containing non-encapsulated lipid) will be ingested after a standardized breakfast, and subsequently satiety and food intake will be measured.
  Arms: Placebo yoghurt

SUMMARY:
This study evaluates the ability of encapsulation of orally applied lipids in a yoghurt snack to modify ad libitum food intake and satiety, without GI symptoms. Every subject receives two treatments (active, and placebo) on two different days, following a randomized cross-over design.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25-30 kg/m2
* Voluntary participation

Exclusion Criteria:

* Milk (-protein or lactose)- allergy/intolerance
* History of serious GI complaints/surgeries
* Pregnancy, lactation
* Excessive alcohol consumption (>20 per week)
* Abnormal eating behaviour
* Intention to stop smoking
* Reported unexplained weight loss or gain in the month prior to screening
* Self-admitted HIV-positive state

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
ad libitum food intake | 2 hours after yoghurt snack
  t=0: standardized breakfast, t=90 minutes: yoghurt, t=210 minutes: ad libitum food intake

SECONDARY OUTCOMES:
Satiety feelings | Up to 3.5 hours on each of the 2 test days.
  Every 15-30 min, 5 attributes will be measured on a Visual Analogue Scale
occurrence and severity of GI symptoms | Up to 3.5 hours on each of the 2 test days.
  Every 15-30 min, 4 attributes will be measured on a Visual Analogue Scale

CONTACTS AND LOCATIONS:
Overall Officials: Adrian AM Masclee, Prof., Principal Investigator — azM/UM
Locations (1):
- Maastricht University, Maastricht, Netherlands

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-29): https://cdn.clinicaltrials.gov/large-docs/97/NCT03025997/Prot_SAP_000.pdf